CLINICAL TRIAL: NCT02998541
Title: A Phase 3, Multi-center, Randomized, Double-Masked Study to Evaluate the Clinical Efficacy and Safety of SHP640 (PVP-Iodine 0.6% and Dexamethasone 0.1%) Ophthalmic Suspension Compared to PVP-Iodine and Placebo in the Treatment of Adenoviral Conjunctivitis
Brief Title: Treatment of Adenoviral Conjunctivitis With SHP640 Compared to Povidone-iodine (PVP-I) and Placebo
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision, unrelated to safety
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP640-301; 2016-002439-14 (EudraCT Number)
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Adenoviral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SHP640 (Experimental): Participants will receive one drop of SHP640 (0.1 percent [%] dexamethasone and 0.6% PVP-I) ophthalmic suspension in each eye 4 times daily (QID) for 7 days.
  Interventions: Drug: SHP640
- PVP-I 0.6% (Active Comparator): Participants will receive one drop of 0.6% PVP-I ophthalmic solution in each eye QID for 7 days.
  Interventions: Drug: PVP-I 0.6%
- Placebo (Placebo Comparator): Participants will receive one drop of placebo ophthalmic solution in each eye QID for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SHP640 — Participants will receive one drop of SHP640 (0.1 % dexamethasone and 0.6% PVP-I) ophthalmic suspension in each eye QID (with a minimum of 2 hours between doses) for 7 days.
  Other Names: FST-100
  Arms: SHP640
Drug: PVP-I 0.6% — Participants will receive one drop of PVP-I ophthalmic solution in each eye QID (with a minimum of 2 hours between doses) for 7 days.
  Arms: PVP-I 0.6%
Other: Placebo — Participants will receive one drop of placebo ophthalmic solution in each eye QID (with a minimum of 2 hours between doses) for 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if an investigational treatment is effective compared with placebo and PVP-Iodine in the treatment of adults and children with adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions (by the parent(s), guardian, or legally authorized representative, if applicable).
* Ability to voluntarily provide written, signed, and dated (personally or via a parent(s), guardian, or legally authorized representative(s) informed consent (and assent, if applicable) to participate in the study.
* Participants of any age at Visit 1 (Note: participants lesser than (<) 3 months of age at Visit 1 must have been full-term, i.e. greater than or equal to (>=) 37 weeks gestational age at birth).
* Meet at least 1 of the 2 criteria below:

  a) Have a positive AdenoPlus test at Visit 1 in at least 1 eye. b) Have at least 2 of the following 5 criteria, based upon medical history and examination: i.Symptoms within the past 7 days consistent with acute upper respiratory tract infection (eg. sore throat, cough, rhinorrhea, etc).

ii. Contact within the past 7 days with family members or other individuals with recent onset of symptoms consistent with conjunctivitis iii. Acute onset within the past 4 days of one or more of the following ocular symptoms: burning/irritation, foreign body sensation, light sensitivity.

iv. Enlarged periauricular lymph node(s). v. Presence of follicles on tarsal conjunctiva. Note:If the participant only meets Inclusion Criterion (a positive AdenoPlus test in at least 1 eye), then the same eye must meet the mentioned below Inclusion Criterion.

* Have a clinical diagnosis of suspected adenoviral conjunctivitis in at least 1 eye confirmed by the presence of the following minimal clinical signs and symptoms in that same eye:

  1. Report presence of signs and/or symptoms of adenoviral conjunctivitis for lesser than or equal to (<=) 4 days prior to Visit 1
  2. Bulbar conjunctival injection: a grade of >= 1 (mild) on a 0-4 Bulbar Conjunctival Injection Scale.
  3. Watery conjunctival discharge: a grade of >= 1 (mild) on a 0-3 Watery Conjunctival Discharge Scale
* Be willing to discontinue contact lens wear for the duration of the study.
* Have a Best Corrected Visual Acuity (BCVA) of 0.60 logMAR or better in each eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. BCVA will be assessed by an age appropriate method in accordance with the AAP Policy Statement for Visual System Assessment in Infants, Children, and Young Adults by Pediatricians (Donahue and Baker 2016; American Academy of Pediatrics 2016).The policy statement recommends formal vision screening can begin at 3 years of age. VA measurements for children under the age of 3 will be done at the discretion of the investigator.
* If not done, child should be able to fixate on and follow a moving object, except participants <2 months of age who have not yet developed this ability. Participants <2 months will be enrolled at the discretion of the investigator.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Exclusion Criteria:

* Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments, per investigator's discretion.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may make the participants unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Have known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.
* Prior enrollment in a FST-100 or SHP640 clinical study.
* Participants who are employees, or immediate family members of employees (who are directly related to study conduct), at the investigational site.
* Have a history of ocular surgical intervention within <= 6 months prior to Visit 1 or planned for the period of the study.
* Have a pre-planned overnight hospitalization during the period of the study.
* Have presence of any intraocular, corneal, or conjunctival ocular inflammation (eg, uveitis, iritis, ulcerative keratitis, chronic blepharoconjunctivitis), other than adenoviral conjunctivitis.
* Have presence of corneal subepithelial infiltrates at Visit 1.
* Have active or history of ocular herpes.
* Have at enrollment or within <= 30 days of Visit 1, a clinical presentation more consistent with the diagnosis of non-infectious conjunctivitis (except presumed seasonal/perennial allergic conjunctivitis), or non-adenoviral ocular infection (e.g. bacterial, fungal, acanthamoebal, or other parasitic).

Note:history or concomitant presence of presumed seasonal or perennial allergic conjunctivitis signs/symptoms is not exclusionary.

* Neonates or infants (i.e. participants less than 12 months of age) who have suspected or confirmed (based on the result of any test conducted prior to screening) conjunctivitis of gonococcal, chlamydial, herpetic or chemical origin.
* Neonates or infants (i.e. participants less than 12 months of age) whose birth mothers had any sexually transmitted disease within 1 month of delivery or any history of genital herpes.
* Presence of nasolacrimal duct obstruction at Visit 1 (Day 1).
* Presence of any significant ophthalmic condition (e.g. Retinopathy of Prematurity, congenital cataract, congenital glaucoma) or other congenital disorder with ophthalmic involvement that could affect study variables.
* Be a known intraocular pressure (IOP) steroid responder, have a known history or current diagnosis of glaucoma, or be a glaucoma suspect.
* Have any known clinically significant optic nerve defects.
* Have a history of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome; presence of corneal epithelial defect or any significant corneal opacity at Visit 1.
* Presence of significant, active condition in the posterior segment which requires invasive treatment (e.g. intravitreal treatment with VEGF inhibitors or corticosteroids) and may progress during the study participation period.
* Have used any topical ocular or systemic anti-vials or antibiotics within <= 7 days of enrollment.
* Have used any topical ocular Non-steroidal Anti-inflammataory Drugs (NSAIDs) within <= 1 day of enrollment.
* Have used any topical ophthalmic steroids in the last <= 14 days.
* Have used any systemic corticosteroid agents within <= 14 days of Day 1. Stable (initiated >= 30 days prior to enrollment) use of inhaled and nasal corticosteroids is allowed, given no anticipated change in dose for the duration of the study. Topical dermal steroids are allowed except in the peri-ocular area.
* Have used non-corticosteroid immunosuppressive agents within <= 14 days of Day 1.
* Have used any topical ophthalmic products, including tear substitutes, and over-the-counter preparations such as lid scrubs, within 2 hours of Visit 1 and be unable to discontinue all topical ophthalmic products for the duration of the study. Use of hot or cold compresses is also not permitted during the study.
* Have any significant ocular disease (eg, Sjogren's syndrome) or any uncontrolled systemic disease or debilitating disease (eg, cardiovascular disease, hypertension, sexually transmitted diseases/infections, diabetes or cystic fibrosis), that may affect the study parameters, per the investigator's discretion.
* Any known history of immunodeficiency disorder or known active conditions predisposing to immunodeficiency, such as human immunodeficiency virus, hepatitis B or C, evidence of active hepatitis A (antihepatitis A virus immunoglobulin M), or organ or bone marrow transplantation.
* Within 30 days prior to the first dose of investigational product:

  1. Have used an investigational product or device, or
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (130):
- United States (68):
  - Arizona Eye Center, Chandler, Arizona
  - Midwestern University Eye Institute, Glendale, Arizona
  - M&M Eye Institute, Prescott, Arizona
  - Walman Eye Center, Sun City, Arizona
  - Milton M. Hom, OD, FAAO, Azusa, California
  - Mark B. Kislinger, MD, PhD, Inc., Glendora, California
  - Inland Eye Specialists, Hemet, California
  - Lakeside Vision Center, Irvine, California
  - Loma Linda University, Loma Linda, California
  - Eye Physicians of Long Beach, Long Beach, California
  - Oxford Optical, Los Angeles, California
  - Macy Eye Center, Los Angeles, California
  - Shultz Chang Vision, Northridge, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Arch Health Partners, Poway, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - The Eye Associates, Bradenton, Florida
  - South Florida Vision Associates, LLC, Fort Lauderdale, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Lorites Medical Group, Miami, Florida
  - Pediatric & Adult Research Center, LLC, Orlando, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Andrew Gardner Logan, MD / dba Logan Ophthalmic Research, LLC, Tamarac, Florida
  - Eye Care Centers Management, Inc., Morrow, Georgia
  - Jackson Eye, Lake Villa, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - MediSphere Medical Research Center, an AMR affiliate, Evansville, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - Koffler Vision Group, Lexington, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - Senior Health Services, Louisville, Kentucky
  - Baker, Carl W, Paducah, Kentucky
  - Lakeview Vision - Gretna, Gretna, Louisiana
  - Haik Humble Eye Center, West Monroe, Louisiana
  - Eye Center Northeast, Bangor, Maine
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Shire Call Center, Lexington, Massachusetts
  - Clinical Eye Research of Boston, Winchester, Massachusetts
  - The Regents of the University of Michigan, Ann Arbor, Michigan
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - Mercy Research, Springfield, Missouri
  - Nevada Eye Care Professionals, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Oculus Research, Raleigh, North Carolina
  - James Branch, M.D., Winston-Salem, North Carolina
  - Matossian Eye Associates, Doylestown, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - The Eye Center at Southern College of Optometry, Memphis, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Eye Specialty Group, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee
  - Toyos Clinic, Nashville, Tennessee
  - Houston Eye Associates, Houston, Texas
  - Lake Travis Eye & Laser Center, Lakeway, Texas
  - Houston Eye Associates, League City, Texas
  - DCT-Shah Research, LLC dba Discovery Clinical Trials, Mission, Texas
  - R and R Eye Research, LLC., San Antonio, Texas
  - Lone Star Eye Care, P.A., Sugar Land, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - Emerson Clinical Research Institute, LLC, Falls Church, Virginia
  - University of Wisconsin, Madison, Wisconsin
- University of the Sunshine Coast Clinical Trials Centre, Sippy Downs, Queensland, Australia
- Austria (3):
  - Kepler Universitätsklinikum, Linz
  - AKH - Medizinische Universitaet Wien, Vienna
  - Vienna Institute for Research in Ocular Surgery, Vienna
- Canada (3):
  - The Ottawa Hospital - General Campus, University of Ottawa Eye Institute, Ottawa, Ontario
  - University of Waterloo School of Optometry and Vision Science, Waterloo, Ontario
  - McGill University Health Centre/Glen Site / Royal Victoria Hospital, Montreal, Quebec
- Estonia (3):
  - Eye Clinic Dr Kirsta Turman, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (2):
  - CHU Limoges - Hopital Dupuytren, Limoges, Haute Vienne
  - Hopital Necker - Enfants Malades, Paris
- Germany (2):
  - Klinisches Studienzentrum der Augenklinik, Mainz
  - Augenärzte am Franziskus Hospital, Münster
- Hungary (5):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Bugat Pal Korhaz, Gyöngyös, Heves County
  - Debreceni Egyetem, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Csolnoky Ferenc Korhaz, Veszprém
- India (12):
  - L. V. Prasad Eye Institute, Hyderabad, Andhra Pradesh
  - Sankara Eye Hospital, Bangalore, Karnataka
  - Bhagwan Mahaveer Jain Hospital, Bangalore, Karnataka
  - M. S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Sapthagiri Hospital, Bangalore, Karnataka
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - NKP Salve Institute of Medical Sciences, Nagpur, Maharashtra
  - Dr. D. Y. Patil Medical College, Navi Mumbai, Maharashtra
  - PBMA'S H. V. Desai Eye Hospital, Pune, Maharashtra
  - S. P. Medical College & Associated Group of Hospitals, Bikaner, Rajasthan
  - ICARE Eye Hospital and Post Graduate Institute, Noida, Uttar Pradesh
  - Regional Institute of Ophthalmology, Kolkata, West Bengal
- Israel (7):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam MC, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- A.O.U. Policlinico San'Orsola-Malpighi, Bologna, Italy
- Peru (3):
  - Instituto Regional de Oftalmología, La Libertad
  - Macula D&T S.R.L., Lima
  - Oftalmosalud SRL., Lima
- Poland (5):
  - Szpital Specjalistyczny nr 1, Bytom
  - Centrum Medyczne UNO-MED, Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - Centrum Medyczne Uno-Med (Private Practice), Tarnów
  - Retina Sp. z o.o., Warsaw
- South Africa (4):
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Into Research, Pretoria, Gauteng
  - Pretoria Eye Institute Research Foundation, Pretoria, Gauteng
  - Nelson R Mandela School of Medicine Ophthalmology Department, Durban, KwaZulu-Natal
- Spain (10):
  - Instituto Oftalmológico Fernández-Vega, Oviedo, Principality of Asturias
  - Complejo Asistencial Universitario de Burgos, Burgos
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Clinica Oftalmologia Gil Piña, Huelva
  - Clinica Rementeria, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Cartuja Vision, Seville
  - FISABIO-Oftalmología Médica, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Manchester Royal Eye Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 97 sites in 15 countries between 27 March 2017 (first participant enrolled) to 13 May 2019 (last participant completed).
Pre-assignment Details: A total of 219 participants were randomized and 196 completed the study. Among which 219 were included in intent-to-treat (ITT) population, 217 in safety population, 83 in modified intent-to treat (mITT) population. Two participants were included in ITT population but not in safety population.
Groups:
- SHP640: Participants administered one drop of SHP640 (0.1 percent [%] dexamethasone and 0.6% PVP-I) ophthalmic suspension in each eye 4 times daily (QID) for 7 days.
- PVP-I 0.6%: Participants administered one drop of 0.6% PVP-I ophthalmic solution in each eye QID for 7 days.
- Placebo: Participants administered one drop of placebo ophthalmic solution in each eye QID for 7 days.
Period: Overall Study
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Started | 86 | 90 | 43
Completed | 78 | 81 | 37
Not Completed | 8 | 9 | 6
Not completed — Adverse Event | 4 | 5 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population consisted of all screened participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | SHP640 | PVP-I 0.6% | Placebo | Total
Number analyzed (Participants) | 86 | 90 | 43 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (19.56) | 42.7 (21.43) | 43.4 (23.67) | 42.3 (21.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 24 | 117
  Male | 40 | 43 | 19 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 16 | 10 | 49
  Not Hispanic or Latino | 63 | 73 | 31 | 167
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 14 | 11 | 5 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 11 | 5 | 25
  White | 62 | 64 | 30 | 156
  More than one race | 0 | 0 | 3 | 3
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Resolution Among Who Received SHP640 or Placebo on Day 6
Description: Clinical resolution of adenoviral conjunctivitis was defined as the absence (score=0) of bulbar conjunctival injection and watery conjunctival discharge in the study eye. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her cell culture-immunofluorescence assay (CC-IFA) results at baseline. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). Higher score represent worse symptoms for both scores. Data analysis was performed in SHP640 and placebo reporting groups only but not in PVP-I 0.6%.
Time Frame: Day 6
Population: Modified Intent to Treat (mITT) population consisted of a subset of the ITT population who received at least one dose of investigational product (IP) and had a positive CC-IFA adenovirus test at baseline in the study eye. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 32 | 0 | 14
Participants | 3 | 0 | 1

2. Secondary Outcome: Number of Participants With Clinical Resolution Among Who Received SHP640 or Povidone-Iodine (PVP-I) on Day 6
Description: Clinical resolution of adenoviral conjunctivitis was defined as the absence (score=0) of bulbar conjunctival injection and watery conjunctival discharge in the study eye. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). Higher score represent worse symptoms for both scores. Data analysis was performed in SHP640 and PVP-I 0.6% reporting groups only but not in placebo.
Time Frame: Day 6
Population: mITT population consisted of a subset of the ITT population who received at least one dose of IP and had a positive CC-IFA adenovirus test at baseline in the study eye. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 32 | 28 | 0
Participants | 3 | 1 | 0

3. Secondary Outcome: Number of Participants With Clinical Resolution Among Who Received Povidone-Iodine (PVP-I) or Placebo on Day 6
Description: Clinical resolution of adenoviral conjunctivitis was defined as the absence (score=0) of bulbar conjunctival injection and watery conjunctival discharge in the study eye. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). Higher score represent worse symptoms for both scores. Data analysis was performed in PVP-I 0.6% and placebo reporting groups only but not in SHP640.
Time Frame: Day 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 28 | 14
Participants | 0 | 1 | 1

4. Secondary Outcome: Number of Participants With Adenoviral Eradication Among Who Received Povidone-Iodine (PVP-I) or Placebo on Day 3
Description: Adenoviral eradication for the study eye was defined as negative Cell Culture- Immunofluorescence Assay (CC-IFA) in that eye. CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Data analysis was performed in PVP-I 0.6% and placebo reporting groups only but not in SHP640.
Time Frame: Day 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 27 | 15
Participants | 0 | 8 | 2

5. Secondary Outcome: Number of Participants With Adenoviral Eradication Among Who Received SHP640 or Placebo on Day 6
Description: Adenoviral eradication for the study eye was defined as negative CC-IFA in that eye. CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Data analysis was performed in SHP640 and placebo reporting groups only but not in PVP-I 0.6%.
Time Frame: Day 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 30 | 0 | 14
Participants | 14 | 0 | 7

6. Secondary Outcome: Number of Participants With Adenoviral Eradication Among Who Received SHP640 or Povidone-Iodine (PVP-I) on Day 6
Description: Adenoviral eradication for the study eye was defined as negative CC-IFA in that eye. CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Data analysis was performed in SHP640 and PVP-I 0.6% reporting groups only but not in placebo.
Time Frame: Day 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 30 | 28 | 0
Participants | 14 | 20 | 0

7. Secondary Outcome: Percent Change From Baseline in Adenovirus Viral Titer as Assessed by Quantitative Polymerase Chain Reaction (qPCR) at Day 6 and 8
Description: qPCR test was performed on all CC-IFA positive samples at all visits to determine viral count in the study eye. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Percent (%) change from baseline in adenovirus viral titer as assessed by qPCR was reported.
Time Frame: Day 6 and 8
Population: The study was terminated as the sponsor discontinued the SHP640 clinical development with reason unrelated to safety. Hence, for this outcome measure, the planned data collection and analysis was not performed.
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Adenoviral Eradication on Day 8 and 12/Early Termination (ET)
Description: Adenoviral eradication for the study eye was defined as negative CC-IFA in that eye. CC-IFA for each eye was conducted using conjunctival swab samples collected at each visit to determine the presence of adenovirus. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline.
Time Frame: Day 8 and 12/ET
Population: mITT population consisted of a subset of the ITT population who received at least one dose of IP and had a positive CC-IFA adenovirus test at baseline in the study eye. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specific categories.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 36 | 32 | 15
Participants
  Day 8: number analyzed (Participants) | 28 | 28 | 15
  Day 8 | 20 | 22 | 13
  Day 12/ET: number analyzed (Participants) | 31 | 31 | 14
  Day 12/ET | 28 | 28 | 13

9. Secondary Outcome: Number of Participants With Clinical Resolution on on Day 3, 8 and 12/Early Termination (ET)
Description: Clinical resolution of adenoviral conjunctivitis was defined as the absence (score=0) of bulbar conjunctival injection and watery conjunctival discharge in the study eye. The study eye was defined based on participant's bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline. Bulbar conjunctival injection was assessed based on a 0 (Normal conjunctival vascular pattern)-4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from the validated bulbar redness (VBR) scale. Watery conjunctival discharge was assessed based on a 0-3 scale (0 - None and 3 - Severe: Abundant quantity of watery discharge observed in the lower conjunctival fornix and in the lower lid margin). Higher score represent worse symptoms for both scores.
Time Frame: Day 3, 8 and 12/ET
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 36 | 32 | 15
Participants
  Day 3: number analyzed (Participants) | 34 | 30 | 15
  Day 3 | 0 | 0 | 0
  Day 8: number analyzed (Participants) | 29 | 28 | 15
  Day 8 | 6 | 5 | 3
  Day 12/ET: number analyzed (Participants) | 32 | 31 | 14
  Day 12/ET | 20 | 13 | 8

10. Secondary Outcome: Change From Baseline in Individual Clinical Signs Score at Day 3, 6, 8 and 12/Early Termination (ET)
Description: The Individual clinical signs score (bulbar conjunctival injection and watery conjunctival discharge) in the study were reported. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CCIFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 7
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With at Least 2 Point Reduction From Baseline in the Global Clinical Score at Day 3, 6, 8 and 12/Early Termination (ET)
Description: Global clinical score was the sum of bulbar conjunctival injection and watery conjunctival discharge. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 36 | 32 | 15
Participants
  Day 3: number analyzed (Participants) | 34 | 30 | 15
  Day 3 | 15 | 5 | 7
  Day 6: number analyzed (Participants) | 32 | 28 | 14
  Day 6 | 22 | 20 | 11
  Day 8: number analyzed (Participants) | 29 | 28 | 15
  Day 8 | 24 | 23 | 13
  Day 12/ET: number analyzed (Participants) | 32 | 31 | 14
  Day 12/ET | 30 | 27 | 12

12. Secondary Outcome: Number of Participants With Modified Clinical Resolution on Day 3, 6, 8 and 12/Early Termination (ET)
Description: Modified clinical resolution was defined as a global clinical score of 0 or 1. Global clinical score was the sum of bulbar conjunctival injection and watery conjunctival discharge. The study eyewas defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 7
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Expanded Clinical Resolution on Day 3, 6, 8 and 12/Early Termination (ET)
Description: Expanded clinical resolution was defined as a global clinical score of 0, 1, or 2 with neither injection nor discharge having a score of 2. Global clinical score was the sum of bulbar conjunctival injection and watery conjunctival discharge. The study eye was defined based on participants bulbar conjunctival redness and watery conjunctival discharge scores at baseline as well as his/her CC-IFA results at baseline.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 7
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Status of Cross-over Infection on Day 3, 6, 8 and 12/Early Termination (ET)
Description: Number of participants with status of cross-over infection to a participant's fellow eye. Participants with only 1 infected eye at baseline were reported.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 7
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Time to Clinical Resolution on Day 3, 6, 8 and 12/Early Termination (ET)
Description: Time to clinical resolution were reported based on the assessments in the study eye.
Time Frame: Day 3, 6, 8 and 12/ET
Population: as for outcome 7
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Event (SAEs) of SHP640
Description: An Adverse Event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A SAE was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, is an important medical event. Any AE that occured after the first dose of IP instillation was considered a TEAE.
Time Frame: From start of the study up to Day 14
Population: Safety Population consisted of all participants who received at least one dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 86 | 90 | 41
Participants
  Treatment-Emergent Adverse Events | 23 | 28 | 10
  Serious Adverse Event | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of the study up to Day 14
Description: Safety Population consisted of all participants who received at least one dose of IP.
Groups:
- SHP640: Participants received one drop of SHP640 (0.1 percent [%] dexamethasone and 0.6% PVP-I) ophthalmic suspension in each eye 4 times daily (QID) for 7 days.
- PVP-I 0.6%: Participants received one drop of PVP-I ophthalmic solution in each eye QID (with a minimum of 2 hours between doses) for 7 days.
- Placebo: Participants received one drop of placebo ophthalmic solution in each eye QID (with a minimum of 2 hours between doses) for 7 days.
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/90 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/90 | 0/41
Other Adverse Events (participants affected / at risk) | 12/86 | 8/90 | 1/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP640 (N=86) | PVP-I 0.6% (N=90) | Placebo (N=41)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP640 (N=86) | PVP-I 0.6% (N=90) | Placebo (N=41)
Instillation site pain (General disorders) | 12 (12) | 8 (8) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated as the sponsor discontinued the SHP640 clinical development with reason unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (5):
  • Study Protocol: Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT02998541/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT02998541/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT02998541/Prot_002.pdf
  • Study Protocol: Amendment 3 (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT02998541/Prot_003.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02998541/SAP_004.pdf